CLINICAL TRIAL: NCT00147680
Title: Prospective, Non-randomised Phase 2 Clinical Trial of Carboplatin Plus Paclitaxel With Sequential Radical Pelvic Radiotherapy for Uterine Serous Papillary Cancer
Brief Title: Uterine Papillary Serous Cancer (UPSC) Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Responsible Party: Prof Andreas Obermair, Queensland Centre for Gynaecological Cancer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPSC - 001
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Uterine Cancer
Keywords: Uterine Papillary Serous Carcinoma (UPSC)
MeSH Terms: conditions — Uterine Neoplasms | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin

SUMMARY:
This study will be an open, non-randomised, clinical phase 2 trial, which will involve 30 women diagnosed with uterine papillary serous cancer. The researchers will investigate the effect of four cycles of paclitaxel/carboplatin, followed by whole pelvic external beam radiotherapy to a standard pelvis field (50.4 Gy) with or without a para-aortic boost with respect to the safety and efficacy of treatment, and patterns of recurrence.

DETAILED DESCRIPTION:
Trial Objectives:

* To assess the safety and efficacy of the combination of Paclitaxel and Carboplatin +/- pelvic radiotherapy in the treatment of UPSC.
* To observe the patterns of recurrence following the administration of the combination of Paclitaxel and Carboplatin +/- pelvic radiotherapy in the treatment of UPSC.
* To assess the QOL, overall survival and disease free survival.

Treatment

Surgery: Total abdominal hysterectomy, bilateral salpingo-oophorectomy, +/- pelvic and aortic node sampling, omentectomy, peritoneal cytology.

Chemotherapy: Chemotherapy commences at the surgeon's and the medical oncologist's discretion and the time between surgery and start of chemotherapy will be recorded. One treatment cycle consists of 3 weeks.

Paclitaxel and Carboplatin will be administered as follows:

Day 1:

* Diphenhydramine 50 mg IV or po or phenergan 12.5 - 25 mg IV
* Cimetidine 300 mg or ranitidine 50 mg IV
* Dexamethasone 20 mg IV
* Paclitaxel 175 mg/m2
* Carboplatin AUC 6

Day 22: Repeat the cycle. This is Day 1 of the second cycle.

Day 43: Repeat the cycle. This is Day 1 of the third cycle.

Day 64: Repeat the cycle. This is Day 1 of the fourth cycle.

Day 85: After the fourth cycle of chemotherapy patients

Patients with stage 4 disease will continue with chemotherapy for a total of 6 cycles.

Patients with surgical stage 1b to 3c disease will receive whole pelvis external beam radiotherapy (50.4 Gy RD over 5 and a half weeks +/- paraaortic boost +/- vaginal vault brachytherapy boost). Radiotherapy will start 4 to 6 weeks after commencement of chemotherapy when the haematological count has recovered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed UPSC at surgical stage 1b to 4 disease. The serous-papillary component of the specimen must be at least 30 percent. Patients with surgical stage 1a disease should not be enrolled.
* Females aged >= 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Patients may not have received any prior chemotherapy regimens for UPSC.
* Patients must have adequate bone marrow, renal, hepatic and neurologic function.
* Patients must be informed of the investigational nature of the study and sign an informed consent form.
* Patients with previous malignancy are eligible only if the patient has been disease-free for >= 5 years.

Exclusion Criteria:

* Patients with pre-existing >= grade 2 neurotoxicity.
* Patients with uncontrolled hypertension, (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg) or uncontrolled cardiac arrhythmia or diabetes mellitus
* Patients with a history of other malignancy within the last 5 years that could affect the diagnosis or assessment of UPSC.
* Patients who have a history of serious cardiac disease that is not adequately controlled are not allowed. Patients with documented myocardial infarction within 6 months preceding study entry; congestive heart failure; unstable angina; a clinically significant pericardial effusion; or arrhythmias are also ineligible.
* Patients with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
* Serious medical or psychiatric illnesses that would prevent informed consent. Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
* Patients with prior significant allergic reactions to drugs containing cremophor, such as cyclosporine, or vitamin K are not eligible. A significant reaction may be defined as, but is not limited to, the description of grade >= 3 allergic reactions using the Common Toxicity Criteria (CTC). Patients with known hypersensitivity to paclitaxel, carboplatin or Cremophor EL.
* Patients who have received prior whole pelvis radiotherapy.
* Patients with uncontrolled pelvic inflammatory disease that would contraindicate pelvic radiotherapy.
* Patients who are pregnant or breast-feeding.
* Patients receiving other investigational therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety and efficacy of the combination of paclitaxel and carboplatin plus/minus (+/-) pelvic radiotherapy in the treatment of UPSC
To observe the patterns of recurrence following the administration of the combination of paclitaxel and carboplatin +/- pelvic radiotherapy in the treatment of UPSC

SECONDARY OUTCOMES:
To assess the quality of life (QOL), overall survival and disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Principal Investigator — QCGC
Locations (2):
- Australia (2):
  - QCGC, Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Public Hospital, South Brisbane, Queensland